CLINICAL TRIAL: NCT04170543
Title: A Phase 2b Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Efficacy and Safety of MEDI3506 in Subjects With Diabetic Kidney Disease
Brief Title: A Phase 2b Diabetic Kidney Disease Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9183C00001
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized to receive MEDI3506 or placebo as follows:
  Group 1: MEDI3506 Dose 1. Group 2: MEDI3506 Dose 2. Group 3: MEDI3506 Dose 3 Group 4: MEDI3506 Dose 4 Group 5: Placebo (volume matched) All subjects will receive Dapa from Day 85 to Day 168.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study in which MEDI3506 and placebo. Neither the subject nor any of the investigator or sponsor staff who are involved in the treatment or clinical evaluation of the subjects will be aware of the treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): MEDI3506 Dose 1 plus Dapagliflozin (Day 85 to Day 168).
  Interventions: Drug: MEDI3506; Drug: Dapagliflozin
- Group 2 (Experimental): MEDI3506 Dose 2 plus Dapagliflozin (Day 85 to Day 168).
  Interventions: Drug: MEDI3506; Drug: Dapagliflozin
- Group 3 (Experimental): MEDI3506 Dose 3 plus Dapagliflozin (Day 85 to Day 168).
  Interventions: Drug: MEDI3506; Drug: Dapagliflozin
- Group 4 (Experimental): MEDI3506 Dose 4 plus Dapagliflozin (Day 85 to Day 168).
  Interventions: Drug: MEDI3506; Drug: Dapagliflozin
- Group 5 (Placebo Comparator): Placebo (volume matched) plus Dapagliflozin (Day 85 to Day 168).
  Interventions: Drug: Placebo; Drug: Dapagliflozin

INTERVENTIONS:
Drug: MEDI3506 — Dose 1, Dose 2, Dose 3, Dose 4
  Arms: Group 1; Group 2; Group 3; Group 4
Drug: Placebo — Placebo
  Arms: Group 5
Drug: Dapagliflozin — Dapagliflozin 10 mg

SUMMARY:
A Phase 2b Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Efficacy and Safety of MEDI3506 in Subjects with Diabetic Kidney Disease

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy, safety, PK, and immunogenicity of MEDI3506 on top of standard of care, including angiotensin-converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs) and dapagliflozin in adult subjects with diabetic kidney disease, defined as subjects with type 2 diabetes mellitus (T2DM) and an estimated glomerular filtration rate (eGFR) of 25-75 mL/min/1.73 m2 with a UACR in the range of 100-3000 mg/g, who meet all eligibility criteria. Approximately 565 subjects, among multiple countries will be randomized to MEDI3506 dose 1, 2, 3 or dose 4, or placebo during a treatment period of 24 weeks. All subjects will receive Dapagliflozin daily, as administered orally from Day 85 to Day 168. The primary objective is to evaluate the effect of MEDI3506 on albuminuria in subjects with DKD. Secondary objectives include evaluating safety, PK and the incidence of ADA during the treatment period.

ELIGIBILITY:
Key Inclusion Criteria

1. Adult men or women ≥ 18 years of age.
2. Diabetic kidney disease DKD defined as:

   1. diagnosis of T2DM
   2. eGFR 25-75 mL/min/1.73 m2
   3. UACR 100-3000 mg albumin/g creatinine
3. BP ≤ 150/100 mmHg
4. Stable dose of ACEi or ARB Key Exclusion Criteria

1. Serum potassium > 5.5 mmol/L 2. Significant hepatic disease 3. Hemoglobin A1c > 10.5 % 4. B-type natriuretic peptide level > 200 pg/mL 5. History of clinically significant heart disease 6. Anticipated dialysis or renal transplantation within 1 year 7. History of underlying condition that predisposes the subject to infections 8. Significant infection (viral, bacterial, or fungal) 9. Amputation due to peripheral artery disease 10. Subjects with a positive diagnostic nucleic acid test for SARS-CoV-2 11. Pregnancy, breastfeeding or intention to become pregnant during the course of the study, 12. Any other medical condition or clinically relevant abnormal findings in physical examination, laboratory results, or electrocardiogram (ECG) during screening that, in the opinion of the investigator, may compromise the safety of the subject in the study, reduce the subject's ability to participate in the study, or interfere with evaluation of the investigational product

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (85):
- United States (45):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Alhambra, California
  - Research Site, Glendale, California
  - Research Site, Granada Hills, California
  - Research Site, Huntington Park, California
  - Research Site, Northridge, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Dimas, California
  - Research Site, Vacaville, California
  - Research Site, Fleming Island, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Manhattan, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Flint, Michigan
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Berlin, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Maumee, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Cypress, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, San Antonio, Texas
  - Research Site, St. George, Utah
  - Research Site, Burke, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Caba
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Pergamino
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, San Luis
  - Research Site, San Nicolás
  - Research Site, San Vicente
- Canada (6):
  - Research Site, Calgary, Alberta
  - Research Site, Red Deer, Alberta
  - Research Site, Brampton, Ontario
  - Research Site, Concord, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Toronto, Ontario
- Chile (4):
  - Research Site, Concepción
  - Research Site, Ñuñoa
  - Research Site, Santiago
  - Research Site, Victoria
- Japan (10):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Ise-shi
  - Research Site, Kisarazu-shi
  - Research Site, Koshigaya-shi
  - Research Site, Nagano
  - Research Site, Nagoya
  - Research Site, Nishinomiya-Shi
  - Research Site, Osaka
  - Research Site, Sayama-Shi
- Research Site, Piura, Peru
- South Korea (7):
  - Research Site, Gangnam-Gu
  - Research Site, Goyang-si
  - Research Site, Jongno-gu
  - Research Site, Seongbuk-Gu
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles.For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Hofherr A, Maki-Petaja K, Selvarajah V, Grice D, Bartesaghi S, Jimenez E, Pecoits-Filho R, Heerspink HJL. Inhibition of IL-33 in Diabetic Kidney Disease: A Randomized, Placebo-Controlled Phase 2b Trial. J Am Soc Nephrol. 2025 Dec 5. doi: 10.1681/ASN.0000000966. Online ahead of print. No abstract available. PMID 41563367
- [Derived] Hofherr A, Liarte Marin E, Musial B, Seth A, Slidel T, Conway J, Baker D, Hansen PBL, Challis B, Bartesaghi S, Bhat M, Pecoits-Filho R, Tu X, Selvarajah V, Woollard K, Heerspink HJL. Inhibition of Interleukin-33 to Reduce Glomerular Endothelial Inflammation in Diabetic Kidney Disease. Kidney Int Rep. 2024 Mar 18;9(6):1876-1891. doi: 10.1016/j.ekir.2024.03.009. eCollection 2024 Jun. PMID 38899206
- See also: D9183C00001_Redacted_CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9183C00001&attachmentIdentifier=c48c8549-14e6-4641-847e-190626b58aeb&fileName=D9183C00001_Redacted_CSP.pdf&versionIdentifier=
- See also: D9183C00001_Redacted_CSR_Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9183C00001&attachmentIdentifier=95604464-a5a6-49a2-854e-e4c573fd0ea2&fileName=D9183C00001_Redacted_CSR_Synopsis.pdf&versionIdentifier=
- See also: D9183C00001_Redacted_SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9183C00001&attachmentIdentifier=f76d1b4f-a37b-4ee1-8117-3091685b8166&fileName=D9183C00001_Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The following data were excluded from this analysis:
  * Data from patients enrolled in Phase 2a of the study: This phase was discontinued due to the COVID-19 pandemic.
  * Data from patients enrolled at a site that was discovered to not follow Good Clinical Practice (GCP) guidelines.
  * Data from patients not treated.
Groups:
- Placebo: Participants were randomized to receive Placebo
- MEDI3506 30 mg: Participants were randomized to receive tozorakimab 30 mg
- MEDI3506 60 mg: Participants were randomized to receive tozorakimab 60 mg
- MEDI3506 120 mg: Participants were randomized to receive tozorakimab 120 mg
- MEDI3506 300 mg: Participants were randomized to receive tozorakimab 300 mg
Period: Overall Study
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Started | 147 | 96 | 101 | 95 | 160
Completed | 99 | 70 | 70 | 68 | 120
Not Completed | 48 | 26 | 31 | 27 | 40
Not completed — Death | 1 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 3 | 3 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 13 | 6 | 5 | 4 | 9
Not completed — Not able to transition to phase 2b | 8 | 0 | 10 | 0 | 6
Not completed — Enrolled in Site with GCP Breach | 6 | 1 | 2 | 2 | 4
Not completed — Not Treated | 0 | 0 | 0 | 0 | 2
Not completed — (CRF) | 16 | 15 | 12 | 17 | 17
Not completed — Due to COVID-19 Pandemic | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg | Total
Number analyzed (Participants) | 133 | 95 | 89 | 93 | 148 | 558
Age, Continuous [Mean (Standard Deviation); unit: years] — The following patients are excluded from reporting:
  1. patients not treated
  2. patients included in Phase 2a who did not have the opportunity to switch to Phase 2b
  3. patients enrolled in the site with GCP breach
  years | 66.7 (9.7) | 67.1 (9.8) | 67.2 (10.1) | 66.6 (9.7) | 65.9 (10.1) | 66.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 46 | 33 | 23 | 24 | 43 | 169
  Sex: Male | 87 | 62 | 66 | 69 | 105 | 389
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 61 | 62 | 31 | 53 | 81 | 288
  Ethnicity: Not Hispanic or Latino | 72 | 33 | 58 | 40 | 67 | 270
  Ethnicity: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 2 | 5 | 0 | 1 | 4 | 12
  Race: Asian | 29 | 15 | 24 | 17 | 29 | 114
  Race: Native Hawaiian or Other Pacific Islander | 1 | 1 | 3 | 1 | 2 | 8
  Race: Black or African American | 16 | 6 | 9 | 4 | 13 | 48
  Race: White | 81 | 68 | 53 | 66 | 96 | 364
  Race: More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Race: Unknown or Not Reported | 3 | 0 | 0 | 4 | 4 | 11
Region of Enrollment [Number; unit: Participants] — The following patients are excluded from reporting:
  1. patients not treated
  2. patients included in Phase 2a who did not have the opportunity to switch to Phase 2b
  3. patients enrolled in the site with GCP breach
  Participants
    Argentina | 20 | 28 | 12 | 28 | 25 | 113
    Canada | 4 | 2 | 7 | 2 | 6 | 21
    Chile | 13 | 12 | 2 | 9 | 17 | 53
    Japan | 20 | 11 | 15 | 11 | 18 | 75
    Korea, Republic of; South Korea | 4 | 3 | 2 | 3 | 3 | 15
    Peru | 0 | 3 | 0 | 0 | 4 | 7
    United States | 72 | 36 | 51 | 40 | 75 | 274

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Day 169 (Week 24) in UACR - Per Protocol Population
Description: UACR values are collected as triplicates at baseline and at each CSP planned visit. For each triplicate, the UACR are averaged with geometric mean.
  Baseline is defined as the geometric mean of UACR measurements prior to first dose of study treatment.
  For the intercurrent events, if a subject is lost to follow-up (EOT), discontinues treatment due to AE, or uses prohibited medication, the UACR data are treated as missing on or after the event and no imputation is performed.
  The LS means of percent change and difference in percent change, corresponding 90% confidence intervals are calculated based on a mixed model with repeated measures (MMRM) of log (UACR post-baseline/UACR baseline) as the response, adjusting for fixed effects of treatment, visit, and treatment-by-visit interaction, SGLT2i, region (Japan or ROW), baseline log UACR, and baseline log UACR-by-visit interaction.
  The MMRM includes UACR values at protocol specified visits from baseline up to Day 169.
Time Frame: From baseline to Day 169
Population: Per Protocol Population:
  All randomized participants who received any study drug and did not violate any relevant important protocol deviations affecting the primary efficacy endpoint.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change from baseline
Groups:
- Placebo: Participants received Placebo
- MEDI3506 30 mg: Participants received tozorakimab 30 mg
- MEDI3506 60 mg: Participants received tozorakimab 60 mg
- MEDI3506 120 mg: Participants received tozorakimab 120 mg
- MEDI3506 300 mg: Participants received tozorakimab 300 mg
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 103 | 81 | 78 | 72 | 131
Percentage change from baseline | -14.82 [-27.05 to -0.53] | -17.25 [-30.69 to -1.19] | -31.45 [-42.54 to -18.21] | -29.70 [-41.61 to -15.37] | -20.96 [-31.32 to -9.04]
Statistical Analysis 1: Comparison: Placebo vs MEDI3506 30 mg; Test type: Other; p = 0.8338, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -2.85, 90% CI 2-sided [-22.61 to 21.94] — MEDI3506 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI3506 60 mg; Test type: Other; p = 0.1169, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -19.52, 90% CI 2-sided [-35.92 to 1.07] — MEDI3506 60 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI3506 120 mg; Test type: Other; p = 0.1774, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -17.47, 90% CI 2-sided [-34.71 to 4.32] — MEDI3506 120 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs MEDI3506 300 mg; Test type: Other; p = 0.5379, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -7.22, 90% CI 2-sided [-24.05 to 13.35]

2. Secondary Outcome: Percent Change From Baseline to Day 85 (Week 12) in UACR - Per Protocol Population
Description: as for outcome 1
Time Frame: From baseline to Day 85
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 103 | 81 | 78 | 72 | 131
Percentage change from baseline | 21.60 [7.39 to 37.70] | 5.77 [-8.00 to 21.60] | -9.66 [-21.46 to 3.91] | -0.53 [-14.10 to 15.18] | 2.69 [-8.32 to 15.01]
Statistical Analysis 1: Comparison: Placebo vs MEDI3506 30 mg; Test type: Other; p = 0.1929, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -13.02, 90% CI 2-sided [-27.08 to 3.75] — MEDI3506 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI3506 60 mg; Test type: Other; p = 0.0062, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -25.71, 90% CI 2-sided [-37.83 to -11.22] — MEDI3506 60 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI3506 120 mg; Test type: Other; p = 0.0705, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -18.20, 90% CI 2-sided [-31.86 to -1.81] — MEDI3506 120 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs MEDI3506 300 mg; Test type: Other; p = 0.0764, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -15.56, 90% CI 2-sided [-27.82 to -1.21]

3. Secondary Outcome: Percent Change From Day 85 (Week 12) to Day 169 (Week 24) in UACR - Per Protocol Population
Description: UACR values are collected as triplicates at baseline and at each CSP planned visit. For each triplicate, the UACR are averaged with geometric mean.
  Baseline is defined as the geometric mean of UACR measurements prior to first dose of study treatment.
  For the intercurrent events, if a subject is lost to follow-up (EOT), discontinues treatment due to AE, or uses prohibited medication, the UACR data are treated as missing on or after the event and no imputation is performed.
  The LS means of percent change and difference in percent change, corresponding 90% confidence intervals are calculated based on a mixed model with repeated measures (MMRM) of log (UACR post-baseline/UACR baseline) as the response, adjusting for fixed effects of treatment, visit, and treatment-by-visit interaction, SGLT2i, region (Japan or ROW), baseline log UACR, and baseline log UACR-by-visit interaction.
  The MMRM includes UACR values at protocol specified visits from Day 85 up to Day 169.
Time Frame: From Day 85 to Day 169
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 103 | 81 | 78 | 72 | 131
Percentage change from baseline | -23.26 [-32.77 to -12.39] | -17.69 [-29.17 to -4.36] | -20.87 [-31.70 to -8.32] | -25.87 [-36.49 to -13.47] | -19.21 [-28.28 to -9]
Statistical Analysis 1: Comparison: Placebo vs MEDI3506 30 mg; Test type: Other; p = 0.5474, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = 7.25, 90% CI 2-sided [-11.45 to 29.88] — MEDI3506 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI3506 60 mg; Test type: Other; p = 0.7920, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = 3.11, 90% CI 2-sided [-14.83 to 24.82] — MEDI3506 60 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI3506 120 mg; Test type: Other; p = 0.7711, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -3.40, 90% CI 2-sided [-20.59 to 17.51] — MEDI3506 120 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs MEDI3506 300 mg; Test type: Other; p = 0.6163, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = 5.27, 90% CI 2-sided [-11.08 to 24.62]

4. Secondary Outcome: Proportion of Subjects With Reduction in UACR at Day 169 (Week 24) - Per Protocol Population
Description: UACR values are collected as triplicates at baseline and at each CSP planned visit. For each triplicate, the UACR are averaged with geometric mean.
  Baseline is defined as the geometric mean of UACR measurements prior to first dose of study treatment.
  Only participants with values at Baseline and Day 169 are included.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 97 | 73 | 74 | 67 | 123
Participants
  UACR reduction > 30% | 43 | 34 | 28 | 38 | 59
  UACR reduction > 40% | 33 | 23 | 23 | 29 | 45
  UACR reduction > 50% | 22 | 17 | 19 | 23 | 35

5. Secondary Outcome: Percent Change From Baseline to Day 169 (Week 24) in UACR - Full Analysis Population
Description: as for outcome 1
Time Frame: From baseline to Day 169
Population: Full Analysis Population:
  All randomized participants who received any study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 133 | 95 | 89 | 93 | 148
Percentage change from baseline | -15.82 [-27.33 to -2.49] | -13.77 [-27.25 to 2.20] | -28.98 [-40.20 to -15.64] | -30.94 [-41.93 to -17.86] | -21.19 [-31.29 to -9.59]
Statistical Analysis 1: Comparison: Placebo vs MEDI3506 30 mg; Test type: Other; p = 0.8537, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = 2.43, 90% CI 2-sided [-17.35 to 26.95] — MEDI3506 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI3506 60 mg; Test type: Other; p = 0.1989, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -15.63, 90% CI 2-sided [-32.14 to 4.89] — MEDI3506 60 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI3506 120 mg; Test type: Other; p = 0.1346, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -17.96, 90% CI 2-sided [-34.01 to 1.99] — MEDI3506 120 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs MEDI3506 300 mg; Test type: Other; p = 0.5683, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -6.38, 90% CI 2-sided [-22.59 to 13.23]

6. Secondary Outcome: Percent Change From Baseline to Day 85 (Week 12) in UACR - Full Analysis Population
Description: as for outcome 1
Time Frame: From baseline to Day 85
Population: Full Analysis Population:
  All randomized participants who received any study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change from baseline
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 133 | 95 | 89 | 93 | 148
Percentage change from baseline | 16.86 [3.59 to 31.83] | 7.59 [-6.16 to 23.35] | -7.23 [-19.29 to 6.63] | -5.03 [-17.55 to 9.39] | 1.35 [-9.52 to 13.53]
Statistical Analysis 1: Comparison: Placebo vs MEDI3506 30 mg; Test type: Other; p = 0.4226, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -7.93, 90% CI 2-sided [-22.30 to 9.10] — MEDI3506 30 mg - Placebo
Statistical Analysis 2: Comparison: Placebo vs MEDI3506 60 mg; Test type: Other; p = 0.0287, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -20.61, 90% CI 2-sided [-33.25 to -5.58] — MEDI3506 60 mg - Placebo
Statistical Analysis 3: Comparison: Placebo vs MEDI3506 120 mg; Test type: Other; p = 0.0498, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -18.73, 90% CI 2-sided [-31.70 to -3.30] — MEDI3506 120 mg - Placebo
Statistical Analysis 4: Comparison: Placebo vs MEDI3506 300 mg; Test type: Other; p = 0.1236, MMRM — Unadjusted two-sided p-value; LS Mean Difference in Percent Change = -13.27, 90% CI 2-sided [-25.51 to 0.98]

7. Secondary Outcome: Proportion of Subjects With Reduction in UACR at Day 169 (Week 24) - Full Analysis Population
Description: as for outcome 4
Time Frame: Baseline and Day 169
Population: Full Analysis Population:
  All randomized participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 108 | 80 | 78 | 77 | 130
Participants
  UACR reduction > 30% | 49 | 36 | 28 | 41 | 62
  UACR reduction > 40% | 37 | 25 | 23 | 32 | 48
  UACR reduction > 50% | 26 | 18 | 19 | 26 | 38

8. Secondary Outcome: Immunogenicity of MEDI3506 - PK Analysis Population
Description: ADA prevalence: number of participants ADA positive (ADA+) at baseline and/or post-baseline.
  Treatment-induced ADA+: ADA not detected or missing at baseline and at least one post-baseline ADA+.
  Treatment-boosted ADA+: ADA+ at baseline and baseline titre is boosted by ≥ 4-fold increase at ≥ 1 post-baseline time point.
  Treatment-emergent ADA+ (TE-ADA + or ADA incidence): Treatment-induced ADA+ OR and Treatment-boosted ADA+.
Time Frame: Day 1 to Day 230
Population: PK Analysis Population:
  All subjects who are randomized and receive any study drug who have at least one detectable MEDI3506 serum concentration measurement post-treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 127 | 92 | 86 | 90 | 146
Participants
  Treatment-induced ADA+ | 1 | 6 | 10 | 12 | 12
  Treatment-boosted ADA+ | 0 | 1 | 0 | 0 | 2
  Treatment-emergent ADA+ (Treatment-induced ADA+ or Treatment-boosted ADA+) | 1 | 7 | 10 | 12 | 14

9. Other Pre Specified Outcome: Plasma Concentration of MEDI3506 - PK Analysis Population
Description: MEDI3506/Tozorakimab serum concentrations were measured using a validated assay method.
Time Frame: Day 1, Day 29, Day 85 and Day 169
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 7 | 94 | 88 | 92 | 147
ng/mL
  Day 1 | 0.01063 (418.9) | 0.005232 (38.16) | 0.005261 (33.33) | 0.005111 (12.30) | 0.005443 (79.38)
  Day 29 | 0.01983 (533.3) | 0.2185 (110.3) | 0.4454 (144.4) | 0.7036 (119.7) | 1.884 (64.34)
  Day 85 | 0.02898 (711.3) | 0.2754 (155.6) | 0.4701 (140.1) | 0.9547 (103.2) | 2.326 (80.10)
  Day 169 | 0.02435 (919.4) | 0.2495 (132.2) | 0.4231 (188.4) | 0.7027 (200.1) | 2.402 (91.04)

10. Secondary Outcome: Asymptomatic Participants Tested Positive for COVID-19 During the Study - Safety Analysis Population
Description: Participants were tested for COVID-19 during the course of the study. Descriptive analysis of asymptomatic participants tested positive for COVID-19 during the study.
Time Frame: Day 1 to Day 230
Population: Safety Analysis Population:
  All randomized participants who received any study drug.
  Subset of participants tested positive for COVID-19 during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 83 | 58 | 53 | 56 | 73
Participants | 79 | 54 | 50 | 53 | 70

11. Secondary Outcome: Treatment-emergent Adverse Events and Treatment-emergent Serious Adverse Events Among COVID-19 Positive Participants - Safety Analysis Population
Description: For participants tested positive for COVID-19 during the intervention and follow-up periods, this analysis provides:
  * the number and proportion of subjects with any treatment-emergent adverse event
  * the number and proportion of subjects with any treatment-emergent serious adverse event
Time Frame: Day 1 to Day 230
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
Number analyzed (Participants) | 83 | 58 | 53 | 56 | 73
Participants
  Any adverse event | 47 | 35 | 23 | 30 | 40
  Any serious adverse event | 11 | 9 | 1 | 6 | 3

ADVERSE EVENTS:
Time Frame: Day 1 to Day 230
Arm/Group | Placebo | MEDI3506 30 mg | MEDI3506 60 mg | MEDI3506 120 mg | MEDI3506 300 mg
All-Cause Mortality (participants affected / at risk) | 1/133 | 1/95 | 1/89 | 1/93 | 1/148
Serious Adverse Events (participants affected / at risk) | 15/133 | 14/95 | 5/89 | 12/93 | 11/148
Other Adverse Events (participants affected / at risk) | 62/133 | 55/95 | 39/89 | 48/93 | 74/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=133) | MEDI3506 30 mg (N=95) | MEDI3506 60 mg (N=89) | MEDI3506 120 mg (N=93) | MEDI3506 300 mg (N=148)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=133) | MEDI3506 30 mg (N=95) | MEDI3506 60 mg (N=89) | MEDI3506 120 mg (N=93) | MEDI3506 300 mg (N=148)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 6 (6) | 3 (3) | 3 (3) | 4 (4) | 5 (5)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (4) | 4 (4) | 0 (0) | 3 (3)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chemical burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 1 (1) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Coagulation test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulse absent (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous pressure jugular increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (7) | 5 (5) | 3 (3) | 9 (10)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 8 (12) | 0 (0) | 2 (2) | 2 (2)
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 2 (2) | 3 (3) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejaculation failure (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile size reduced (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic dermopathy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Onychogryphosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 6 (6) | 1 (1) | 7 (7) | 7 (7)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Corneal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (6) | 3 (3) | 4 (4)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Granuloma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (5)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 4 (4) | 1 (1) | 2 (2) | 6 (7)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
41 randomized participants were excluded from analysis populations in order to avoid heterogeneity in the data (bias, etc.) :

* 2 participants did not received any IP
* 24 participants were enrolled in phase 2a without having the possibility to be enrolled in phase 2b
* 15 participants were randomized in a site with GCP breach (inability to confirm the validity of the data reported)

These 41 participants are excluded from Baseline characteristics (558 participants).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04170543/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04170543/SAP_001.pdf